CLINICAL TRIAL: NCT02689232
Title: TEG (Thromboelastography) Based Versus Conventional Coagulation Parameters Based Correction of Coagulopathy in Non Variceal Bleed: An Open Label Randomized Controlled Trial.
Brief Title: TEG (Thromboelastography) Based Versus Conventional Coagulation Parameters Based Correction of Coagulopathy in Non Variceal Bleed.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ILBS-Variceal Bleed-001
Record Dates: First submitted 2016-02-13; First posted 2016-02-23 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-02

CONDITIONS: Non Variceal Bleed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thromboelastography (TEG) level (Experimental)
  Interventions: Biological: Fresh Frozen Plasma; Biological: Platelets Concentrate; Biological: Cryo Precitipitate
- Coagulation Profile (Active Comparator)
  Interventions: Biological: Fresh Frozen Plasma; Biological: Platelets Concentrate; Biological: Cryo Precitipitate

INTERVENTIONS:
Biological: Fresh Frozen Plasma
Biological: Platelets Concentrate
Biological: Cryo Precitipitate

SUMMARY:
All patients with non variceal bleed who are admitted under the Department of Hepatology at Institute of Liver and Biliary Sciences, who meet the inclusion criteria and who provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18
* All patient with Non Variceal bleed (INR>1.8 and platelets<50000)
* Hist logical or imaging proven liver cirrhosis.

Exclusion Criteria:

1. Variceal Bleed,
2. Pregnancy.,
3. Patients on anticoagulation
4. Patients who refused to participate in the study
5. Post EVL ulcer bleed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2018-03-03 (Actual); Study Completion 2018-03-03 (Actual)

PRIMARY OUTCOMES:
Amount of FFP (Fresh Frozen Plasma) transfusion in both groups | 42 days

SECONDARY OUTCOMES:
Number of patients with bleed in both groups | 5 days
Incidence of TRALI (Transfusion associated lung injury) and TACO ( Transfusion associated circulatory overload) in both the groups. | 42 days
Early mortality ( <6 weeks) and late mortality (> 6 weeks) in both the groups. | 42 days
Amount of blood products (Platelet and cryo and Red Blood Cells)transfused in both the groups. | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr Juned Ahmad, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (2):
- India (2):
  - Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi
  - Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kumar M, Ahmad J, Maiwall R, Choudhury A, Bajpai M, Mitra LG, Saluja V, Mohan Agarwal P, Bihari C, Shasthry SM, Jindal A, Bhardwaj A, Kumar G, Sarin SK. Thromboelastography-Guided Blood Component Use in Patients With Cirrhosis With Nonvariceal Bleeding: A Randomized Controlled Trial. Hepatology. 2020 Jan;71(1):235-246. doi: 10.1002/hep.30794. Epub 2019 Aug 27. PMID 31148204